CLINICAL TRIAL: NCT01574391
Title: A COMPARISON STUDY OF TWO DIFFERENT TECHNIQUES FOR IDENTIFYING THE EPIDURAL SPACE IN PARTURIENTS IN LABOUR: A PILOT PROSPECTIVE RANDOMIZED STUDY.
Brief Title: A Comparison Study Of Two Different Techniques For Identifying The Epidural Space In Parturients In Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Maternity Hospital, Ireland (Other)
Responsible Party: Principal Investigator, DR ROGER MCMORROW, DR ROGER MCMORROW, National Maternity Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMHEPI-12
Record Dates: First submitted 2012-04-08; First posted 2012-04-10 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Labouring Parturients Requiring/Requesting Epidural Analgesia as Part of Their Peri-partum Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPIDRUM (Active Comparator): EPIDRUM DEVICE IS USED TO SITE THE EPIDURALS IN THE PATIENTS RANDOMISED TO THIS ARM
  Interventions: Device: Epidrum
- Control (No Intervention): This arm is the control where normal technique is used

INTERVENTIONS:
Device: Epidrum — Epidrum is used
  Other Names: Epidrum is the trade name of the device manufactured by Exmore Plastics Uk
  Arms: EPIDRUM

SUMMARY:
The purpose of this study is to determine whether the use of the Epidrum device to identify the epidural space in labouring parturients reduces morbidity, when compared to standard loss of resistance techniques.

ELIGIBILITY:
Inclusion Criteria:

* Parturients receiving epidural analgesia for labour

Exclusion Criteria:

* parturients that withold consent
* parturients less than 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
RATE OF OCCURRENCE OF DURAL PUNCTURE | FIRST 48 HRS

SECONDARY OUTCOMES:
RATE OF EPIDURAL BLOOD PATCH | I MONTH AFTER LAST PATIENT RECRUITED
RATE OF EPIDURAL FAILURE REQUIRING RE-SITING OF CATHETER | 24 HOURS
RATE OF FAILURE IN IDENTIFYING EPIDURAL SPACE REQUIRING CHANGE OF OPERATOR | 24

CONTACTS AND LOCATIONS:
Locations (1):
- National Maternity Hospital, Dublin, Co Dublin, Ireland